CLINICAL TRIAL: NCT05749315
Title: Comparative Effects of Play Based Therapy and Functional Communication Training in Speech-language Delayed Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muniba001-09
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Speech, Language Developmental Delay From Hearing Loss
Keywords: Play based therapy; Functional communication training
MeSH Terms: conditions — Speech | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A Speech Language Delayed Children
  Interventions: Other: Play Based Therapy
- Group B (Active Comparator): Group B Speech Language Delayed Children
  Interventions: Other: Functional Communication Training

INTERVENTIONS:
Other: Play Based Therapy — Participants' assessments of SLD will be made using the Portage Guide to Early Education. It will take three months of sessions 5 days a week, lasting 20 to 30 minutes. The individual will be asses through Speech Questionnaire on base line and after 3 months session program. The Progress of both therapies will be seen that which technique is more effective.
  Arms: Group A
Other: Functional Communication Training — Participants' assessments of SLD will be made using the Portage Guide to Early Education. It will take three months of sessions 5 days a week, lasting 20 to 30 minutes. The individual will be asses through Speech Questionnaire on base line and after 3 months session program. The Progress of both therapies will be seen that which technique is more effective.
  Arms: Group B

SUMMARY:
The purpose of this study is to compare the play based therapy and functional communication training in speech-language delayed children 2-6 years old. This study will highlight the most effective intervention or therapy for Speech & Language Delayed Children. The Randomized clinical trial study will be conducted in clinic, sehat medical complex, with children who will have the diagnosis of speech and language delay. These individual will be diagnose by a speech therapist (more than 2 years experience in the field) with PORTAGE guide to early education . A group of children will be given play based therapy and the other group of children will be given functional communication training. Participants' assessments of SLD will be made using the Portage Guide to Early Education. It will take three months of sessions 5 days in a week, lasting 20 to 30 minutes. The Progress of both therapies will be seen and assessed through structured questionnaire that which technique is more effective. The individual will be assess through Speech Questionnaire on base line and after 3 months session program.

DETAILED DESCRIPTION:
Speech is the verbal production of language, whereas language is the conceptual processing of communication. Language includes receptive language (understanding) and expressive language (the ability to convey information, feelings, thoughts, and ideas). Language is commonly thought of in its spoken form, but may also include a visual form, such as American Sign Language. Speech and language delay in children is associated with increased difficulty with reading, writing, attention, and socialization. In children not meeting the expected milestones for speech and language, a comprehensive developmental evaluation is essential, because atypical language development can be a secondary characteristic of other physical and developmental problems that may first manifest as language problems.

ELIGIBILITY:
Inclusion Criteria:

* Participants with comorbidity of behavioral disorder, Autism & ADHD

Exclusion Criteria:

* Patient with comorbidity of syndromes ( downs syndrome, treacher Collin syndrome, hunter syndrome , Williams Syndrome, kabuki syndrome etc )

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Speech Questionnaire | Change from baseline at 3rd Month
  The Speech Questionnaire: an Assessment of Functional Language Ability. International Rehabilitation Medicine.

CONTACTS AND LOCATIONS:
Overall Officials: Momina Mehmood, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan